CLINICAL TRIAL: NCT00539838
Title: A Randomised, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy and Safety of Two Doses of Ocrelizumab in Patients With Active Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate Two Doses of Ocrelizumab in Patients With Active Systemic Lupus Erythematosus (BEGIN)
Acronym: BEGIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated prematurely when the decision was made that ocrelizumab was not likely to benefit this patient population.
Sponsor: Genentech, Inc. (Industry)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT4071g; WA20499
Record Dates: First submitted 2007-10-03; First posted 2007-10-05 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Prednisone; Azathioprine; Mycophenolic Acid; Methotrexate; Methylprednisolone; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Ocrelizumab 1000 mg (Experimental): Ocrelizumab was administered i.v. at a dose on Days 1 and 15, followed by 1000 mg i.v. at Week 16 and then every 16 weeks
  Interventions: Drug: Prednisone; Drug: Immunosuppressive regime (azathioprine, mycophenolate mofetil or methotrexate); Drug: Methylprednisolone; Drug: Ocrelizumab
- Ocrelizumab 400 mg (Experimental): Ocrelizumab was administered at a dose 400 mg i.v. on Days 1 and 15, followed by 400 mg i.v. at Week 16 and then every 16 weeks
  Interventions: Drug: Prednisone; Drug: Immunosuppressive regime (azathioprine, mycophenolate mofetil or methotrexate); Drug: Methylprednisolone; Drug: Ocrelizumab
- Placebo (Placebo Comparator): Placebo infusions were administered on Days 1 and 15, followed by placebo infusion at Week 16 and then every 16 weeks
  Interventions: Drug: Immunosuppressive regime (azathioprine, mycophenolate mofetil or methotrexate); Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Oral repeating dose
  Arms: Ocrelizumab 1000 mg; Ocrelizumab 400 mg
Drug: Immunosuppressive regime (azathioprine, mycophenolate mofetil or methotrexate) — Oral repeating dose
Drug: Methylprednisolone — Intravenous repeating dose
  Arms: Ocrelizumab 1000 mg; Ocrelizumab 400 mg
Drug: Ocrelizumab — Intravenous repeating dose
  Arms: Ocrelizumab 1000 mg; Ocrelizumab 400 mg
Drug: Placebo — Intravenous repeating dose
  Arms: Placebo

SUMMARY:
This is a Phase III, randomized, double blind, placebo-controlled, multicenter, parallel-group study to evaluate the efficacy and safety of ocrelizumab compared to placebo when combined with a single stable background immunosuppressive medication and a corticosteroid regimen in patients with moderately to severely active systemic lupus erythematosus, who do not have moderate to severe glomerulonephritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years or above at the time of screening
* Diagnosis of SLE
* Active disease at screening

Exclusion Criteria:

* Presence of active moderate to severe glomerulonephritis
* Currently active retinitis, poorly controlled seizure disorder, acute confusional state, myelitis, stroke or stroke syndrome, cerebellar ataxia, or dementia
* Lack of peripheral venous access
* Pregnancy or breast feeding mothers
* History of severe allergic or anaphylactic reactions to humanized, chimeric or murine monoclonal antibodies or i.v. immunoglobulin
* Known severe chronic pulmonary disease
* Evidence of significant or uncontrolled concomitant diseases in any organ system not related to SLE, which, in the investigator's opinion, would impair patient participation
* Concomitant condition which has required treatment with systemic corticosteroid (excluding topical or inhaled) at any time in the 52 weeks prior to screening
* Known HIV or chronic active Hepatitis B or chronic active Hepatitis C infection
* Known active infection of any kind (but excluding fungal infection of nail beds or oral thrush which has resolved before Day 1) within 30 days prior to Day 1. In addition, any major episode of infection requiring hospitalization or treatment with intravenous anti-infectives in the 30 days prior to Day 1 or oral anti-infectives in the 14 days prior to Day 1
* History of serious recurrent or chronic infection
* History of cancer (except basal cell carcinoma of the skin that has been excised and cured)
* History of alcohol or drug abuse in the 52 weeks prior to screening
* Major surgery in the 4 weeks prior to screening excluding diagnostic surgery
* Previous treatment with CAMPATH-1H
* Previous treatment with a BAFF directed treatment in the 12 months prior to screening
* Previous treatment with a B-cell targeted therapy other than one directed at BAFF
* Treatment with any investigational agent, other than those above, in the 28 days prior to screening or five half-lives of the investigational drug (whichever is longer)
* Receipt of any live vaccine in the 6 weeks prior to Day 1
* Intolerance or contraindication to oral or i.v. corticosteroids
* Treatment with a second immunosuppressive or immunomodulatory drug in the 8 weeks prior to Day 1
* Prednisone dose of ≥ 0.7 mg/kg/day (or equivalent) for > 7 of the previous 30 days prior to screening
* Treatment with cyclophosphamide or a calcineurin inhibitor in the 12 weeks prior to screening
* Positive hepatitis BsAg or hepatitis C serology. Patients who are HBsAg negative but HBcAb positive may be enrolled with a negative DNA test

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-12-19 (Actual); Primary Completion 2011-07-12 (Actual); Study Completion 2011-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorn Drappa, M.D., Ph.D., Study Director — Genentech, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A maximum screening window of 14 days was allowed.
Pre-assignment Details: During the screening period, participants received oral prednisone after the physician's evaluation and scoring of a BILAG questionnaire.
Period: Overall Study
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Started | 12 | 11 | 10
Completed | 5 | 5 | 1
Not Completed | 7 | 6 | 9
Not completed — Fail to return | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 0
Not completed — Death | 0 | 2 | 0
Not completed — Did not cooperate | 1 | 0 | 1
Not completed — Administrative | 4 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ocrelizumab 400 mg | Ocrelizumab 1000 mg | Total
Number analyzed (Participants) | 10 | 11 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (13.82) | 40.2 (8.80) | 36.3 (11.31) | 39.0 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 10 | 30
  Male | 1 | 0 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 4 | 12
  Not Hispanic or Latino | 4 | 9 | 8 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 3 | 8
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 5 | 8 | 7 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Clinical Response (MCR)
Time Frame: Week 48
Population: Evaluation of the primary and some secondary endpoints was to occur at Week 48 with further analyses conducted at Week 96. However, following the early termination of the study, the analysis of the primary and secondary endpoints were not conducted.
Arm/Group | Placebo | Ocrelizumab 400 mg | Ocrelizumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Partial Clinical Response (PCR)
Time Frame: Week 48
Population: as for outcome 1
Arm/Group | Placebo | Ocrelizumab 400 mg | Ocrelizumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Number of Non-responders (NR)
Time Frame: Week 48
Population: as for outcome 1
Arm/Group | Placebo | Ocrelizumab 400 mg | Ocrelizumab 1000 mg
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Who Achieved a BILAG Score of C or Better at Week 24.
Time Frame: Week 24
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Time Adjusted Mean SLEDAI-2K Score
Time Frame: Week 48
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Annualized Flare Rate
Time Frame: Week 48 to Week 96
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Time to First Moderate to Severe Flare
Time Frame: Week 48 to Week 96
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Who Achieved A Major Or Partial Clinical Response At Week 48 (PCR Plus MCR Proportion), Who Did Not Experience A Flare Before Week 96
Time Frame: Week 48 to Week 96
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Who Achieved A MCR At Week 48, Who Did Not Experience A Flare Before Week 72
Time Frame: Week 48 to Week 72
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Achieved A MCR At Week 48, Who Did Not Experience A Flare Before Week 96
Time Frame: Week 48 to Week 96
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change in SF-36 Subscale And Summary Scores From Baseline At Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change In FACIT-Fatigue Assessment From Baseline To Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline In Pain Quality And Impact Of Pain On Daily Function Measured By The Brief Pain Inventory Short Form At Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: The EQ-5D Single Index Utility Score At Week 48
Time Frame: Baseline, Week 48
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 2.5 years
Population: as for outcome 1
Arm/Group | Ocrelizumab 1000 mg | Ocrelizumab 400 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 42 months.
Description: Multiple occurrences of the same adverse event in one individual counted only once
Arm/Group | Placebo | Ocrelizumab 400 mg | Ocrelizumab 1000 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 6/11 | 3/12
Other Adverse Events (participants affected / at risk) | 5/10 | 10/11 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Ocrelizumab 400 mg (N=11) | Ocrelizumab 1000 mg (N=12)
CYTOMEGALOVIRUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CHORIORETINITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMOCYSTIS JIROVECI (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | Ocrelizumab 400 mg (N=11) | Ocrelizumab 1000 mg (N=12)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CYTOMEGALOVIRUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CHORIORETINITIS FUNGAL SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
NAIL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ONYCHOMYCOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECI (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
TINEA CRURIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VAGINITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
TONGUE DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
HEMIANOPIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
POST HERPETIC NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (General disorders) | 0 (0) | 2 (2) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
SWELLING (General disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0)
NODULE ON EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
VITAMIN D DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
MENISCUS LESION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
AMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated before any patients reached the Week 48 visit. Therefore, the safety analysis included all safety data for the 33 randomized patients that were available up to the data cutoff date (22 March 2010)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.